CLINICAL TRIAL: NCT06908720
Title: A Prospective Observational Study for Defining the Role of Optical Super-high Magnification Dermoscopy in the Diagnosis of Skin Tumors
Brief Title: Defining the Role of Optical Super-high Magnification Dermoscopy in the Diagnosis of Skin Tumors
Acronym: OSHMD
Status: Not yet recruiting | Type: Observational
Sponsor: IRCCS Ospedale San Raffaele (Other)
Responsible Party: Principal Investigator, Guida Stefania, Dr. Stefania Guida is a medical doctor, Specialist in Dermatology and Venereology, and holds a PhD in "Clinical and Experimental Medicine." She currently holds the position of researcher at the Clinical Dermatology Unit at HSR, IRCCS Ospedale San Raffaele
Other Study IDs: CET 58-2025 (OSHMD)
Record Dates: First submitted 2025-03-26; First posted 2025-04-03 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-04

CONDITIONS: Skin Cancers
MeSH Terms: conditions — Skin Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
This is a prospective study aimed at evaluating the diagnostic accuracy (compared to histopathological diagnosis) and clinical utility of optical super-high magnification dermoscopy (OSHMD) in detecting and differentiating skin tumors, including both benign and malignant lesions, particularly in nevi/melanoma and basal cell carcinoma, in patients with suspicious lesions at a magnification of 20x. Additionally, the characteristics of skin lesions will be analyzed using OSHMD, and their distribution in skin tumors will be assessed. The agreement between the examiners' evaluations and the concordance between dermoscopic diagnoses at 20x and 400x compared to histopathological diagnosis will also be examined. The hypothesis is that OSHMD could assist in identifying malignancy features, thus improving the diagnostic accuracy of skin tumors and potentially leading to earlier and more precise detection of neoplasms

ELIGIBILITY:
Inclusion Criteria:

* patients who will come to our attention for skin cancer screening with dermoscopy, willing to partecipate to the study

Exclusion Criteria:

* patients aged under 18 year old
* patients unable to understand and signed the onformed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients who will come to our attention for skin cancer screening with dermoscopy, willing to partecipate to the study
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Evaluate the diagnostic accuracy and clinical utility of super-high magnification dermoscopy in the detection and differentiation of skin tumors | from the enrollment to the reaching of 1000 patients or up to 156 weeks
  Accuracy (sensibility and specificity) of dermoscopy 400x for detecting skin tumors (vs histopathological diagnosis)